CLINICAL TRIAL: NCT02008604
Title: Influence of Stroke on the Composition of Intestinal Microbiota (GUTSTROKE)
Brief Title: Influence of Stroke on the Composition of Intestinal Microbiota
Acronym: GUTSTROKE
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Prof. Dr. Ulrich Dirnagl, Experimental Neurology, Charité Berlin, Germany (Unknown); Dr. Christian Meisel, Medical Immunology, Charité Berlin, Germany (Unknown); PD Dr. Andreas Nitsche, Robert-Koch-Institut, Berlin, Germany (Unknown); NeuroCure Clinical Research Center, Charite, Berlin (Other)
Responsible Party: Principal Investigator, Andreas Meisel, Prof. Dr., Charite University, Berlin, Germany
Other Study IDs: GUTSTROKE
Record Dates: First submitted 2013-11-15; First posted 2013-12-11 (Estimated); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Stroke; Transient Ischemic Attack (TIA)
Keywords: ischemia; stroke; transient ischemic attack (TIA); microbiome; microbiota; gut
MeSH Terms: conditions — Stroke; Ischemic Attack, Transient; Ischemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool samples, Blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Stroke patients
- TIA patients: patients with a transient ischemic attack (control group)

SUMMARY:
The aim of the study is to verify the hypothesis that the microbial colonisation of the gut is changed in patients after stroke and that the gut microbiome of severely affected stroke patients differs from that of patients with only a short disruption of blood circulation in the brain (transient ischemic attack, TIA). For this, the composition of gut microbiota in stool samples will be analyzed by 454 pyrosequencing. Further, the correlation of stroke-associated changes in the microbiome with immunological parameters will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* age: 18 and older
* ischemic cerebral infarction within the last 40 hours, anterior circulation infarct (ACA, MCA) and/or posterior circulation infarct (PCA, BA) of any severity
* patient consent or consent by a legal representative
* NIHSS > or =9 (stroke patients)
* NIHSS < 1 (for TIA patients)

Exclusion Criteria:

* intracranial hemorrhage
* preexisting dysphagia
* signs of infection upon admission (clinical/paraclinical)
* existing antibiotic therapy upon admission or within the last 2 weeks before admission
* mechanical ventilation upon admission
* participation in an interventional therapy study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients at the rescue center, the Stroke Unit and the neurological intensive care unit of the Charité University hospital
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
composition of intestinal microbiome | change between day 1, day 4, day 7, day 14 after stroke
  The composition of the intestinal metagenome / microbiome will be determined by analyzing the 16S rRNA by 454 Pyrosequencing.

SECONDARY OUTCOMES:
test of correlation between most changed group of bacteria with changes in immunological parameters (HLA-DR) | days 1, 4, 7 after stroke
  Analysis of correlation between changes in microbiome (most changed group of bacteria, e.g. lactobacilli) with changes in immunological parameters (e.g. HLA-DR, IL-6, IL-10, CD4-lymphocytes from blood samples).

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Meisel, Prof. Dr., Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charite Universitätsmedizin Berlin, Berlin, Germany